CLINICAL TRIAL: NCT04301401
Title: Assessment of Changes in Vaginal Microbiota Profiles Before and After Vaginal Urogynecologic Surgery
Acronym: VAGIBIOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NIMAO/2019-01/LA-01
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Gynecological Surgery
Keywords: Microbiota; vagina; prolapse; transvaginal surgery; surgical site infection
MeSH Terms: conditions — Prolapse; Surgical Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients being evaluated for changes in microbiota (Experimental): Patients being evaluated for changes in vaginal microbiota following transvaginal surgery.
  Interventions: Other: Vaginal swabs; Other: Stool samples; Other: Urine samples

INTERVENTIONS:
Other: Vaginal swabs — On the day of the surgical intervention, vaginal swabs will be taken at various stages of surgery: before vaginal disinfection/draping, directly after disinfection/draping, 1 hour after disinfection, 6 weeks after surgery and 12 months after surgery.
Other: Stool samples — Stool samples will also be taken (and collected in a pot devoted to coproculture with an airtight opaque bag given to the patient) at the inclusion visit on the day before surgery and also 6 weeks after surgery (in a second pot with an airtight opaque bag given to the patient at the time of being discharged).
Other: Urine samples — Urine samples will also be taken before surgery and 6 weeks after surgery.

SUMMARY:
Several studies have shown interactions between vaginal microbiota and post-surgical evolution. A study conducted by our team showed a tendency for patients with complications to have a greater diversity of vaginal microbiota. The main objective of the proposed study will therefore be to evaluate the vaginal, urinary and digestive microbiota modifications during and after vaginal surgery and to correlate them with the symptoms of the urogynecological sphere.

DETAILED DESCRIPTION:
In gynecological surgery, surgical site infections are a common complication. Gynecological surgery and, more specifically, vaginal surgery leads to a high risk of infection not only due to its " clean-contaminated " nature related to the proximity of the vagina but also due to the use of a transvaginal mesh or suburetal sling. The germs most commonly found at the origin of a surgical site infection are germs forming part of the vaginal flora.

Furthermore, in the field of pelvic organ prolapse surgery, certain specific complications such as mesh retraction and mesh exposure may be related to infection due to bacterial colonisation.

The vaginal ecosystem contains a large quantity of bacteria, the commonest of which are lactobacilli. This ecosystem varies in women depending on their sexuality, hormonal impregnation, tobacco consumption or hygiene.It has been demonstrated that the microbiota can be divided into 7 classes depending on the predominant types of germ. It has also been shown that an imbalance in vaginal flora could be responsible for infections of the upper genital tract, obstetric complications or even the transmission of sexually transmissible diseases.

Several studies have shown interactions between the microbiota and post surgical evolution. A recent study carried out at the Gynecology and Obstetrics department of Nîmes University Hospital (Veit Rubin et al, NAU 2019) also investigated the relationship between vaginal microbiota and the onset of postoperative complications in transvaginal mesh surgery. This retrospective study also found that patients with complications tended to have a greater diversity of microbiota. Furthermore, certain species of bacteria (Veillonella spp) seemed to be commoner in patients with complications. However, this was a low-powered retrospective study with few participants and the results therefore need to be confirmed.

Our hypothesis is that the vaginal microbiota may be modified by a surgical act with a vaginal approach. There are very few studies on vaginal microbiota and so far no studies have evaluated the potential impact of a transvaginal surgery on vaginal microbiota.

Our study may help to better understand the relationship between the vaginal microbiota and the postoperative evolution of patients.These possible modifications in vaginal microbiota might be predictive of the symptomatology of patients benefitting from transvaginal surgery and play a role in the the post-operative evolution of these patients.

ELIGIBILITY:
Inclusion Criteria:

* All Caucasian menopausal women (not taking hormone substitutes)
* Due to undergo transvaginal surgery (as a cure for pelvic organ prolapse or stress urinary incontinence surgery) from the Gynecology departments of Nantes and Nîmes University Hospitals.
* Patients must be covered by a health insurance policy
* Patients must have given written, informed consent.

Exclusion Criteria:

* Patients on recent (<1 month) immunosuppressive therapy,
* Patients with ongoing antibiotic therapy,
* Patients with chronic vaginosis,
* Patients on hormone replacement therapy
* Patients who have had previous transvaginal mesh surgery.
* Patients taking part in another category 1 study for research involving human subjects.
* Patients in an exclusion period determined by another study
* Patients under court custody, guardianship or curatorship
* Patients for whom it has been impossible to give clear information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Menopausal women
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Classes of vaginal flora before surgery | Day 1
  A vaginal swab will be taken before surgery and the sample will be analyzed by DNA sequencing in order to classify the microbiota into community state types.
Classes of vaginal flora 6 weeks after surgery | Day 42
  A vaginal swab will be taken 6 weeks after surgery and the sample will be analyzed by DNA sequencing in order to classify the microbiota into community state types.

SECONDARY OUTCOMES:
Classes of vaginal flora 12 mois after surgery | Month 12
  A vaginal swab will be taken 12 months after surgery and the sample will be analyzed by DNA sequencing in order to classify the microbiota into community state types.
Alphadiversity of vaginal flora before preparation for surgery measured with the Shannon index | Day 1
  A vaginal swab will be taken before any preparation for surgery has begun and the alphadiversity of the microbiota will be measured according to the Shannon index in Taxonomic Operational Units
Betadiversity of vaginal flora before preparation for surgery measured with the Bray-Curtis index | Day 1
  A vaginal swab will be taken before any preparation for surgery has begun and the betadiversity of the microbiota will be measured according to the Bray-Curtis index in Taxonomic Operational Units
Alphadiversity of vaginal flora directly after disinfection and draping, measured with the Shannon index | Day 1
  A vaginal swab will be taken directly after disinfection and draping and the alphadiversity of the microbiota will be measured according to the Shannon index in Taxonomic Operational Units.
Betadiversity of vaginal flora directly after disinfection and draping, measured with the Bray-Curtis index | Day 1
  A vaginal swab will be taken directly after disinfection and draping and the betadiversity of the microbiota will be measured according to the Bray-Curtis index in Taxonomic Operational Units.
Alphadiversity of vaginal flora one hour after disinfection and draping, measured with the Shannon index | Day 1
  A vaginal swab will be taken one hour after disinfection and draping and the alphadiversity of the microbiota will be measured according to the Shannon index in Taxonomic Operational Units.
Betadiversity of vaginal flora one hour after disinfection and draping, measured with the Bray-Curtis index | Day 1
  A vaginal swab will be taken one hour after disinfection and draping and the betadiversity of the microbiota will be measured according to the Bray-Curtis index in Taxonomic Operational Units.
Alphadiversity of vaginal flora six weeks after surgery, measured with the Shannon index | Day 42
  A vaginal swab will be taken six weeks after surgery and the alphadiversity of the microbiota will be measured according to the Shannon index in Taxonomic Operational Units.
Betadiversity of vaginal flora six weeks after surgery, measured with the Bray-Curtis index | Day 42
  A vaginal swab will be taken six weeks after surgery and the betadiversity of the microbiota will be measured according to the Bray-Curtis index in Taxonomic Operational Units.
Alphadiversity of vaginal flora twelve months after surgery, measured with the Shannon index | Month 12
  A vaginal swab will be taken twelve months after surgery and the alphadiversity of the microbiota will be measured according to the Shannon index in Taxonomic Operational Units.
Betadiversity of vaginal flora twelve months after surgery, measured with the Bray-Curtis index | Month 12
  A vaginal swab will be taken twelve months after surgery and the betadiversity of the microbiota will be measured according to the Bray-Curtis index in Taxonomic Operational Units.
Prolapse. Feeling a bulge six weeks after surgery | Day 42
  Yes/No. If present, this will be classified according to the International Continence Society-International Urogynecological Association classification
Prolapse. Feeling a bulge twelve months after surgery | Month 12
  Yes/No. If present, this will be classified according to the International Continence Society-International Urogynecological Association classification
Dyspareunia six weeks after surgery | Day 42
  Yes/no. If present, this will be rated according to the International Continence Society-International Urogynecological Association classification.
Dyspareunia 12 months after surgery | Month 12
  Yes/No. If present, this will be rated according to the International Continence Society-International Urogynecological Association classification.
Pain six weeks after surgery | Day 42
  The patient will be asked to evaluate pain according to a visual analogue scale ranging from 0 (no pain) to 10 (extremely painful).
Pain 12 months after surgery | Month 12
  The patient will be asked to evaluate pain according to a visual analogue scale ranging from 0 (no pain) to 10 (extremely painful).
Urinary incontinence upon effort six weeks after surgery | Day 42
  Yes/No. If present, this will be rated according to the International Continence Society-International Urogynecological Association classification.
Urinary incontinence upon effort 12 months after surgery | Month 12
  Yes/No.If present, this will be classified according to the International Continence Society-International Urogynecological Association classification
Need to urinate urgently six weeks after surgery | Day 42
  Yes/No.If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Need to urinate urgently 12 months after surgery | Month 12
  Yes/No.If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Dysuria 6 weeks after surgery | Day 42
  Yes/No.If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Dysuria 12 months after surgery | Month 12
  Yes/No.If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Constipation 6 weeks after surgery | Day 42
  Yes/No. If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Constipation 12 months after surgery | Month 12
  Yes/No. If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Anal incontinence 6 weeks after surgery | Day 42
  Yes/No. If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Anal incontinence 12 months after surgery | Month 12
  Yes/No. If present, this will be classified according to the International Continence Society-International Urogynecological Association classification.
Presence or absence of complications 6 weeks after surgery | Day 42
  Yes/No. If present, these will be rated according to the Clavien Dindo classification. The Clavien Dindo classification is a scale with grades ranging from 1 to 5 in which Grade 1 = any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside. Grade 5 = death of the patient.
Presence or absence of complications 12 months after surgery | Month 12
  Yes/No. If present, these will be rated according to the Clavien Dindo classification.The Clavien Dindo classification is a scale with grades ranging from 1 to 5 in which Grade 1 = any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside. Grade 5 = death of the patient.
Presence or absence of complications related to a prosthesis 6 weeks after surgery | Day 42
  Yes/No. If present, these will be rated according to the International Continence Society-International Urogynecological Association classification
Presence or absence of complications related to a prosthesis 12 months after surgery | Month 12
  Yes/No. If present, these will be rated according to the International Continence Society-International Urogynecological Association classification.
Presence or absence of infection at the operating site 6 weeks after surgery | Day 42
  Yes/No
Presence or absence of infection at the operating site 12 months after surgery | Month 12
  Yes/No
Urine sample before surgery | Day 1
  A urine sample will be collected from the patient before surgery and stored in a sterile pot at -80° at the Biological resource Centre at Nîmes or Nantes University Hospitals.
Urine sample after vaginal disinfection and surgical draping. | Day 1
  A urine sample will be collected from the patient before surgery but after vaginal disinfection and surgical draping, and stored in a sterile pot at -80° at the Biological resource Centre at Nîmes or Nantes University Hospitals.
Urine sample 6 weeks after surgery six weeks after surgery | Day 42
  A urine sample will be collected from the patient 6 weeks after surgery and stored in a sterile pot at -80° at the Biological resource Centre at Nîmes or Nantes University Hospitals.
Urine sample 12 months after surgery | Month 12
  A urine sample will be collected from the patient 12 months after surgery and stored in a sterile pot at -80° at the Biological resource Centre at Nîmes or Nantes University Hospitals.
Stool sample before surgery | Day 0
  The day before surgery, at the inclusion visit, a stool sample will be collected in a sterile pot and stored at -80° at the Biological resource Centre at Nîmes or Nantes University Hospitals.
Stool sample 6 weeks after surgery | Day 42
  Six weeks after surgery, a stool sample will be collected in a sterile pot and stored at -80° at the Biological resource Centre at Nîmes or Nantes University Hospitals.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Nîmes, Gard, France

REFERENCES:
- [Result] Zhang Y, Allegre L, Salipante F, Morsli M, Thubert T, Lavigne JP, Dunyach-Remy C, de Tayrac R. Impact of surgical field disinfection on vaginal microbiome in transvaginal urogynecological surgery: a prospective cohort study. Antimicrob Resist Infect Control. 2025 Aug 26;14(1):102. doi: 10.1186/s13756-025-01622-6. PMID 40859385